CLINICAL TRIAL: NCT01399086
Title: A Retrospective Study of Fulvestrant in Postmenopausal Patients With Metastatic Breast Cancer in Greece (The 'RESPONSE' Study)
Brief Title: Fulvestrant in Postmenopausal Patients With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CT/10.10
Record Dates: First submitted 2011-05-23; First posted 2011-07-21 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: Cancer; Breast; Metastatic; Hormonotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fulvestrant
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — 250mg on d1,15,29 or 250mg on d1 q28days
  Other Names: Faslodex

SUMMARY:
This is a retrospective chart-review study that will be based on the collection of data from electronical or paper-based medical records with available data on patients who have commenced treatment with fulvestrant after January 1st of 2007. All necessary information for the purposes of the present study will be collected with the use of a paper-Case Record Form.

DETAILED DESCRIPTION:
To date, there are no available data on the use of fulvestrant in the treatment of postmenopausal women with metastatic breast cancer in current clinical practice in Greece. In view of this significant lack of knowledge, we designed this retrospective study in order to evaluate the effectiveness of fulvestrant in real-life settings, by obtaining data regarding the use of fulvestrant in current clinical practice among treating physicians in Greece. This retrospective study aims to address the following questions:

* What is the clinical outcome of fulvestrant treatment in terms of TTP when used in metastatic breast cancer in a real life clinical setting?
* What is the positioning of fulvestrant in the hormone therapy sequencing in metastatic breast cancer in Greece?
* What are the other clinical outcomes (ORR, duration of response, CBR) of fulvestrant treatment in metastatic breast cancer in a real life clinical setting and what is the relation between clinical outcomes and fulvestrant's position in the treatment sequence?
* What is the usual duration of fulvestrant treatment in metastatic breast cancer in the real life clinical setting and which are the reasons for treatment discontinuation?
* Treatment failure with fulvestrant: what is the next step in sequencing according to patients' breast cancer treatment history?

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with ER-positive and/or PgR-positive breast cancer who have failed at least one prior endocrine therapy, either as adjuvant treatment or for the treatment of advanced disease
* Patients who have received treatment with fulvestrant for metastatic breast cancer and have completed/discontinued the treatment regardless of outcome/reason for discontinuation (except for treatment discontinuation for non-clinical reasons)
* Patients who were at postmenopausal status at the time of treatment with fulvestrant

Exclusion Criteria:

* Patients who are currently undergoing treatment with fulvestrant
* Investigators/treating physicians with no available electronical or paper-based medical records

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective chart-review study that will be based on the collection of data from electronical or paper-based medical records with available data on patients that fulfil the following-mentioned eligibility criteria and have initiated therapy with fuvestrant after January 1st of 2007. All necessary information for the purposes of the present study will be collected with the use of a paper-Case Record Form
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Time to Progression | 1 year
  To evaluate the time to progression (TTP) from the initiation of fulvestrant treatment in postmenopausal women with endocrine-positive breast cancer who have failed at least one prior endocrine therapy, either as adjuvant treatment or for the treatment of advanced disease

SECONDARY OUTCOMES:
Objective Response Rate | > 6 months
  To evaluate the objective response rate (ORR), i.e. the rate of both complete and partial response, and to estimate the duration of response while on treatment with fulvestrant
Tumor growth control | >6 months
  To evaluate the clinical benefit rate (CBR), i.e. the rate of both complete and partial response as well as stable disease ≥ 6 months, while on treatment with fulvestrant, where applicable

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (9):
- Greece (9):
  - "Ag.Georgios" General Hospital of Chania, Chania, Crete
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "Agios Savvas" Anticancer Hospital of Athens, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - IASO General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - Theagenion Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki